CLINICAL TRIAL: NCT06904703
Title: Combination of Pericapsular Nerve Group and Lumbar Erector Spinae Plane Blocks for Geriatrics Undergoing Total Hip Arthroplasty Under General Anesthesia: A Randomized Controlled Trial
Brief Title: Pericapsular Nerve Group and Lumbar Erector Spinae Plane Blocks for Geriatrics Undergoing Total Hip Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mai El-saieed Abdelghaffar Hamada, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Management Department, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36265MD311/11/24
Record Dates: First submitted 2025-03-22; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Pericapsular Nerve; Lumbar Erector Spinae Plane Blocks; Geriatrics; Total Hip Arthroplasty; General Anesthesia
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- General anesthesia group (Experimental): Patients will receive general anesthesia.
  Interventions: Drug: General anesthesia
- Erector spinae plane block group (Experimental): Patients will receive general anesthesia and erector spinae plane block.
  Interventions: Drug: Bupivacaine 0.5%
- Pericapsular nerve block group (Experimental): Patients will receive general anesthesia and erector spinae plane block with pericapsular nerve block.
  Interventions: Drug: Bupivacaine 0.5%

INTERVENTIONS:
Drug: General anesthesia — Patients will receive general anesthesia.
  Arms: General anesthesia group
Drug: Bupivacaine 0.5% — Patients will receive general anesthesia and erector spinae plane block.
  Other Names: Erector spinae plane block
  Arms: Erector spinae plane block group
Drug: Bupivacaine 0.5% — Patients will receive general anesthesia and erector spinae plane block with pericapsular nerve block.
  Other Names: Pericapsular nerve block
  Arms: Pericapsular nerve block group

SUMMARY:
This study will be conducted to evaluate the effect of pericapsular nerve group and erector spinae plane block as adjuvants to general anesthesia in geriatrics undergoing total hip arthroplasty.

DETAILED DESCRIPTION:
Total hip arthroplasty is one of the most common major orthopedic procedures to improve a patient's functional status and quality of life. Total hip arthroplasty is one of the most cost-effective and consistently successful surgeries performed in orthopedics and can be associated with significant postoperative pain.

General anesthesia may be considered more versatile and suitable for patients with complex medical histories or those who cannot tolerate spinal anesthesia. However, older patients undergoing hip fracture surgery under general anesthesia may experience a higher risk of postoperative delirium, prolonged sedation, and respiratory complications. Moreover, delayed mobilization is possible, leading to a higher incidence of complications such as deep vein thrombosis and pressure sores.

The target nerves of the hip joint arise from the lumbar plexus (L1-L4), the lumbosacral trunk of the sacral plexus (L4-L5), and the sacral spinal nerves (S1-S4) (7). The femoral nerve, obturator nerve, and the accessory obturator nerve supply the anterior capsule of the hip; the sciatic nerve and the nerve to the quadratus femoris mostly supply the articular branches to the posterior capsule of the hip joint The erector spinae plane block is a novel inter-fascial plane block targets the dorsal and ventral rami of the spinal nerves, is a newer regional anesthetic technique that can be used to provide analgesia for a variety of surgical procedures or to manage acute or chronic pain. This block can potentially provide analgesia to the posterior pelvis potentially safer alternative to epidural or paravertebral techniques, areas often involved in hip fracture pain.

The pericapsular nerve group block targets the articular branches of the femoral and obturator nerves near the hip joint capsule. By blocking these nerves, the pericapsular nerve group block effectively provides analgesia to the hip joint, particular tissues, and proximal femur.

ELIGIBILITY:
Inclusion Criteria:

* Aged >75 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) classification I-III.
* Undergoing total hip arthroplasty under general anesthesia.

Exclusion Criteria:

* Patient refusal.
* Body mass index (BMI) > 30 kg/m2.
* Allergy to local anesthesia drugs.
* Infection at the site of intervention.
* Coagulopathies.
* Preexisting advanced diseases of the kidney or liver.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Mean sevoflurane MAC to achieve bispectral index (BIS) values (45-55) | Intraoperatively
  Sevoflurane will be adjusted to maintain a steady state with a BIS value in the range of 45-55 and will be fixed through the study period

SECONDARY OUTCOMES:
Pain degree | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the Numerical Rating Scale (NRS). NRS (0 represents "no pain" while 10 represents "the worst pain imaginable").Pain intensity will be measured using a 10-point NRS at rest at 2, 4, 8, 12, 18, and 24 hours postoperatively.
Fentanyl consumption. | Intraoperatively
  Additional fentanyl bolus dosages of 1 µg/kg IV will be administered if heart rate or mean arterial blood pressure elevated more than 20% of the baseline (after exclusion of other causes than pain).
Arterial blood pressure | Till the end of surgery (up to 2 hours)
  MAP will be recorded pre-induction of anesthesia, post-induction of anesthesia and before performing of block, and every 15 min till the end of surgery. Intraoperative arterial blood pressure will be assessed. Hypotension (decrease in basal mean arterial blood pressure by 20%) will be treated with IV fluid.
Heart rate | Till the end of surgery (up to 2 hours)
  HR will be recorded pre-induction of anesthesia, post-induction of anesthesia and before performing of block, and every 15 min till the end of surgery.
Total postoperative morphine consumption. | First 24 hours after surgery
  Total postoperative morphine consumption in the first 24h after surgery will be recorded. Rescue analgesia of morphine will be given as 0.05mg/kg bolus if the Numerical Rating Scale (NRS) > 3 to be repeated after 30 min if pain persists until the NRS < 4.
Patient satisfaction | 24 hours after surgery
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied). It will be assessed 24 hours after surgery.
Complications | 24 hours Postoperatively
  Complications such as bradycardia, hypotension, nausea, vomiting, pruritis, respiratory depression will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one yea
Access Criteria: The data will be available upon a reasonable request from the corresponding author